CLINICAL TRIAL: NCT05517525
Title: An Open-label, Phase 1 Study to Evaluate the Pharmacokinetics and Safety of a Single Dose of Brensocatib in Subjects With Normal Hepatic Function and Subjects With Hepatic Impairment
Brief Title: A Study to Evaluate the Pharmacokinetics (PK) and Safety of a Single Dose of Brensocatib in Participants With Normal Hepatic Function and Participants With Hepatic Impairment
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Insmed Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: INS1007-105
Record Dates: First submitted 2022-08-24; First posted 2022-08-26 (Actual); Last update posted 2023-07-19 (Actual); Status verified 2023-07

CONDITIONS: Hepatic Impairment
Keywords: Brensocatib; INS1007
MeSH Terms: interventions — brensocatib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Cohort 1: Brensocatib (Experimental): Healthy participants with normal hepatic function will receive single oral dose of brensocatib on Day 1 under fasted conditions. Healthy participants will be matched within the protocol criteria to one or more participants with hepatic impairment.
  Interventions: Drug: Brensocatib
- Cohort 2: Brensocatib (Experimental): Participants with mild hepatic impairment will receive single oral dose of brensocatib on Day 1 under fasted conditions.
  Interventions: Drug: Brensocatib
- Cohort 3: Brensocatib (Experimental): Participants with moderate hepatic impairment will receive single oral dose of brensocatib on Day 1 under fasted conditions.
  Interventions: Drug: Brensocatib
- Cohort 4: Brensocatib (Experimental): Participants with severe hepatic impairment will receive single oral dose of brensocatib on Day 1 under fasted conditions.
  Interventions: Drug: Brensocatib

INTERVENTIONS:
Drug: Brensocatib — Oral tablet.
  Other Names: INS1007

SUMMARY:
The primary purpose of the study is to compare the PK of a single dose of brensocatib in participants with hepatic impairment to that in matched healthy control participants with normal hepatic function.

ELIGIBILITY:
Inclusion Criteria:

- Has body mass index (BMI) between 18.0 and 35.0 kilogram per square meter (kg/m^2)

Inclusion Criteria for Participants With Hepatic Impairment:

* Clinical diagnosis of chronic hepatic disease, as documented in their medical history of underlying hepatic insufficiency with features of cirrhosis and no acute episodes of illness within 30 days prior to screening, and no significant change in disease status from screening to check-in.
* Hepatic impairment will be classified using the Child-Pugh criteria
* A stable medication regimen, defined as not starting new drug(s) or changing dosage(s) within 30 days prior to study drug administration. Concomitant medications must be approved by the investigator and medical monitor.

Inclusion Criteria for Healthy Matched Control Participants With Normal Hepatic Function:

* In good health, determined by no clinically significant findings from medical history, clinical laboratory evaluations, vital signs measurements, 12-lead electrocardiogram (ECG), and physical examination at screening or check-in, as assessed by the investigator (or designee).
* Matched to hepatically impaired participants in age (±10 years), sex, and BMI (±20%).

Exclusion Criteria:

* History of stomach or intestinal surgery or resection that would potentially alter absorption and/or excretion of orally administered drugs (uncomplicated appendectomy and hernia repair will be allowed; cholecystectomy will not be allowed).
* Positive human immunodeficiency virus (HIV) test
* Administration of a coronavirus disease 2019 (COVID-19) vaccine in the past 30 days prior to dosing.
* Participation in a clinical study involving administration of an investigational drug (new chemical entity) in the past 30 days prior to dosing.
* Use of moderate to strong CYP3A4 inducers or inhibitors within 14 days prior to check-in.
* Have previously completed or withdrawn from this study or any other study investigating brensocatib, and have previously received the IMP.

Exclusion Criteria for Participants With Hepatic Impairment:

* Positive urine drug screen at screening or check-in, unless the result is due to a prescribed medication.
* History of significant immunologic impairment such as transplantation.
* Hepatic encephalopathy Grade ≥2 using Child-Pugh scoring.

Exclusion Criteria for Healthy Matched Control Participants with Normal Hepatic Function

* Positive urine drug screen at screening or check-in.
* Significant history or clinical manifestation of any immunologic, metabolic, allergic, dermatological, hepatic, renal, hematological, pulmonary, cardiovascular, gastrointestinal, neurological, respiratory, endocrine, or psychiatric disorder, as determined by the investigator (or designee).
* Positive hepatitis panel. Participants whose results are compatible with prior immunization are eligible at the discretion of the investigator.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2022-10-04 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-06-01 (Actual)

PRIMARY OUTCOMES:
Area Under the Concentration Time Curve (AUC) | Pre-dose and at multiple timepoints post-dose on Days 1 to 9
  Comparison of the pharmacokinetics of a single dose of brensocatib in participants with hepatic impairment to that in matched healthy control participants with normal hepatic function.

SECONDARY OUTCOMES:
Fraction Unbound (Fu) | Pre-dose and at multiple timepoints post-dose on Days 1 to 9
  Assessment of the plasma protein binding of brensocatib in participants with varying degrees of hepatic function relative to matched healthy control participants with normal hepatic function.
Number of Participants who Experienced at Least one Adverse Event (AE) | From first dose of study drug up to follow up visit (5-7 days after discharge) or early termination (up to Day 17)
  Determination of the safety and tolerability of a single dose of brensocatib in participants with hepatic impairment.

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - USA002, Rialto, California
  - USA003, Orlando, Florida
  - USA001, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Usansky H, Au Yeung S, Li S, Marbury T, Lawitz E, Kayali Z, Stein DS. Pharmacokinetics and Safety of a Single Dose of Brensocatib in Participants with Hepatic Impairment and Matched Participants with Normal Hepatic Functions. Clin Pharmacokinet. 2026 Jan 26. doi: 10.1007/s40262-025-01614-0. Online ahead of print. PMID 41586857